CLINICAL TRIAL: NCT00242151
Title: Prevalence of Delirium in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHN REB 05-0223-AE
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-09

CONDITIONS: Heart Disease
Keywords: Delirium, Confusion, Cardiac Surgery, Organic Brain Injury, Diffusion Weighted Magnetic Resonance Imaging (DW-MRI)
MeSH Terms: conditions — Heart Diseases; Delirium; Confusion

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The objective of this study is to determine prevalence of postoperative delirium and confusion in patients undergoing cardiac surgery. This proposal is a pilot study designed to evaluate effect of cardiac surgery on prevalence of delirium and confusion.

The primary aim is to evaluate prevalence of delirium and confusion in patients undergoing cardiac surgery and to determine risk factors for this condition.

A secondary aim is to evaluate organic brain injury by early postoperative diffusion weighted magnetic resonance imaging (DW-MRI) in patients who develop delirium and confusion.

The hypothesis to be tested is that patients with postoperative delirium and confusion have high incidence of organic brain injury as detected by DW-MRI.

ELIGIBILITY:
Inclusion criteria:

* All patients undergoing cardiac surgery in our institute in 2 year period
* Signed informed consent

Exclusion criteria:

* Past history of transient ischemic attacks, stroke, symptomatic carotid artery disease.
* Past history of psychiatric disorders
* History of alcohol and drug abuse
* History of severe kidney or liver disease (creatinine >2.5mg/dL and bilirubin > 2mg/dL)
* Known contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada